CLINICAL TRIAL: NCT04363333
Title: Impact of Obstructive Sleep Apnea on Covid-19 Outcomes (OSACOVID-19 Study): A Prospective Observational Cohort Study
Brief Title: Obstructive Sleep Apnea & Covid-19 Outcomes
Acronym: OSACOVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Koç University (Other)
Collaborators: Koc Healthcare Istanbul American Hospital, Marmara University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020.140.IRB1.030
Record Dates: First submitted 2020-04-19; First posted 2020-04-27 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: COVID; Obstructive Sleep Apnea; Pneumonia
Keywords: COVID; Obstructive Sleep Apnea; Pneumonia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Probability of OSA: Based on a sleep questionnaire
  Interventions: Diagnostic Test: Home Sleep Apnea Testing or In-hospital Polysomnography
- Low Probability of OSA: Based on a sleep questionnaire
  Interventions: Diagnostic Test: Home Sleep Apnea Testing or In-hospital Polysomnography

INTERVENTIONS:
Diagnostic Test: Home Sleep Apnea Testing or In-hospital Polysomnography — Home Sleep Apnea Testing or In-hospital Polysomnography will be conducted 4 to 6 months after the Covid-19 diagnosis

SUMMARY:
Covid-19 infection is an on-going pandemic with worse diagnosis in adults with comorbid conditions such as hypertension and cardiopulmonary diseases. Obstructive sleep apnea (OSA) is common in those comorbidities and may contribute to worse prognosis for the Covid-19 cases.

DETAILED DESCRIPTION:
The investigators' primary aim is to address the association between the high probability of having OSA and Covid-19 outcomes within 28 days of the hospitalization.

Secondary outcomes will be conducting a polysomnography in cases with high probability of having OSA compared to those with low probability, approx. 4 months after the Covid-19 diagnosis, and re-evaluate the association of the verified OSA diagnosis and severity with the outcomes in the first 4 weeks as well as with the outcomes after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Covid 19 diagnosis
* Ability to read and speak
* Signed informed consent.

Exclusion Criteria:

* Subjects with limited life expectancy due to advanced renal disease or uncontrolled malignancies
* Subjects with alcohol dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Covid-19 diagnosis
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
The rate of clinical improvement | 7 days
  Defined as a decline of 2 categories from admission on a 7-category ordinal scale
The rate of clinical improvement | 14 days
  Defined as a decline of 2 categories from admission on a 7-category ordinal scale
The rate of clinical improvement | 21 days
  Defined as a decline of 2 categories from admission on a 7-category ordinal scale
The rate of clinical improvement | 28 days
  Defined as a decline of 2 categories from admission on a 7-category ordinal scale

SECONDARY OUTCOMES:
Clinical status - improvement | 7, 14, 21, 28 days
  Time to hospital discharge, ICU discharge, weaning from intubation, weaning from supplemental oxygen, incident pneumonia, ARDS, in-hospital mortality
Clinical status - worsening | 7, 14, 21, 28 days
  Defined as an increase in category on a 7-category ordinal scale from admission

OTHER OUTCOMES:
Long-term outcomes | 4-6 months after the initial hospital admission
  Re-analysis of the correlation of obstructive sleep apnea (objectively verified) severity in terms of apnea-hypopnea index and oxygenation levels with the primary and secondary outcomes as described above (the rate of clinical improvement defined as a decline of 2 categories from admission on a 7-category ordinal scale; time to hospital discharge, ICU discharge, weaning from intubation, weaning from supplemental oxygen, incident pneumonia, ARDS, in-hospital mortality as well as with the lung function, CO-diffusion capacity, cardiac function, CT thorax pathologies, biomarkers (cytokines, polymorphisms) and IgG-antibodies after 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yuksel Peker, MD, PhD, Study Chair — Koc University School of Medicine
Locations (3):
- Turkey (Türkiye) (3):
  - Marmara University Hospital, Istanbul, Basibuyuk
  - Koc University, Istanbul
  - Koc Healthcare Istanbul American Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results that will be reported in articles would be available to other researchers by contacting the corresponding authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months after the publications, respectively
Access Criteria: Within 6 months after the publications, respectively, for 5 years

REFERENCES:
- [Derived] Peker Y, Celik Y, Arbatli S, Isik SR, Balcan B, Karatas F, Uzel FI, Tabak L, Cetin B, Baygul A, Ozturk AB, Altug E, Iliaz S, Atasoy C, Kapmaz M, Yazici D, Bayram H, Cetin BD, Caglayan B; OSACOVID-19 Study Collaborators. Effect of High-Risk Obstructive Sleep Apnea on Clinical Outcomes in Adults with Coronavirus Disease 2019: A Multicenter, Prospective, Observational Clinical Trial. Ann Am Thorac Soc. 2021 Sep;18(9):1548-1559. doi: 10.1513/AnnalsATS.202011-1409OC. PMID 33596161